CLINICAL TRIAL: NCT07305272
Title: Evaluation of the Effect of Animated Video-Assisted Nutrition Education on Nutritional Behaviors, Symptom Severity, and Quality of Life in Heart Failure Patients
Brief Title: Evaluation of the Effect of Animated Video-Assisted Nutrition Education on Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Yasemin BOY, Research Assistant, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GOU-2025-RCT-001
Record Dates: First submitted 2025-11-15; First posted 2025-12-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; Nutrition Education; Animation Video; Dietary Behavior; Symptom Severity; Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients will receive animation video-supported nutrition education focusing on balanced diet, sodium restriction, sugar and cholesterol control, and fluid retention prevention. Videos will follow the "5W1H and Symptom" principle. Follow-ups will be at 1 month, 3 months, and 6 months using HF Dietary Behavior Scale, HF Symptom Status Scale, and Minnesota Living with HF Questionnaire.
  Interventions: Behavioral: Animation Video-Supported Nutrition Education
- Control Group (No Intervention): Patients will receive standard care (verbal advice from cardiologists) and will complete the same assessments at baseline, 1 month, 3 months, and 6 months. After study completion, they will also receive access to the animation video education.

INTERVENTIONS:
Behavioral: Animation Video-Supported Nutrition Education — Structured education using animation videos on balanced diet, sodium restriction, sugar/cholesterol control, fluid retention prevention. Videos delivered in hospital and accessible on patients' phones for 6 months with weekly reminders.
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of animation video-supported nutrition education on dietary behaviors, symptom severity, and quality of life in patients with heart failure. A total of 70 patients aged 45-60 years with NYHA class II or III heart failure will be recruited at Tokat Gaziosmanpaşa University Research and Application Hospital Cardiology Clinic. Participants will be randomly assigned to an intervention group, which will receive video-supported nutrition education, or a control group, which will receive standard care. Outcomes will be assessed using the Heart Failure Dietary Behavior Scale, Heart Failure Symptom Status Scale, and Minnesota Living with Heart Failure Questionnaire at baseline, 1 month, 3 months, and 6 months.

DETAILED DESCRIPTION:
This study investigates the effect of animation video-supported nutrition education on dietary behaviors, symptom severity, and quality of life in patients with heart failure (HF). The study will be conducted at Tokat Gaziosmanpaşa University Research and Application Hospital Cardiology Clinic from July 2025 to December 2025. A total of 70 patients aged 45-60 years with NYHA class II or III HF will be included. Patients meeting the inclusion criteria and willing to participate will be randomly assigned to the intervention or control group using a computer-based simple randomization method.

The intervention group will receive a structured nutrition education program delivered through animation videos developed based on clinical guidelines, focusing on balanced nutrition, sodium restriction, sugar and cholesterol control, and fluid retention prevention. Videos will illustrate key concepts using the "5W1H and Symptom" (What, Where, How, When, Why, Symptom) principle. Baseline assessments will include the Heart Failure Dietary Behavior Scale, Heart Failure Symptom Status Scale, Minnesota Living with Heart Failure Questionnaire, and a demographic form. Follow-up assessments will be conducted at 1 month, 3 months, and 6 months.

The control group will receive standard care, including verbal advice from cardiologists. After completion of the study, control group patients will also have access to the animation video education. Data will be analyzed using SPSS v25 with appropriate statistical tests, and linear mixed-effects models will be applied to evaluate group, time, and group-time interaction effects.

ELIGIBILITY:
Inclusion Criteria:

Individuals who have been diagnosed with heart failure at least six months ago,

* Are between the ages of 45-60,
* Are in NYHA stage II or III,
* Have a mobile phone capable of watching videos,
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

Individuals with HF who were included in the study as a sample,

* Patients with fluid restriction under a different protocol (e.g., Chronic Renal Failure),
* Patients with chronic pulmonary disease (e.g., COPD),
* Illiterate,
* Do not own a mobile phone capable of watching videos,
* Have physical or cognitive impairments,
* Have a psychiatric illness,
* Refuse to participate in the study will not be included in the study.
* Patients hospitalized during the study period will be excluded from the study, and their data will not be subject to statistical analysis.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Mean Score on the Heart Failure Dietary Behavior Scale | At baseline, 1 month, 3 months, and 6 months
  Dietary behaviors will be evaluated using the Heart Failure Dietary Behavior Scale, developed by Boy and Enç (2022). The scale consists of 19 items across four subscales: Healthy Habits, Salt Restriction, Sugar Restriction, and Prevention of Fluid Retention. Items are rated on a 4-point Likert scale, yielding a total score range of 19-76. Higher scores indicate better adherence to dietary recommendations. A cutoff score of 46 is used; scores ≥46 indicate adherence to guideline-recommended nutritional behaviors.

SECONDARY OUTCOMES:
Mean Score on the Heart Failure Symptom Status Scale (Symptom Severity) | At baseline, 1 month, 3 months, and 6 months
  Symptom severity will be assessed using the Heart Failure Symptom Status Scale, developed by Heo et al. (2015). This patient-reported outcome measure evaluates the presence, frequency, severity, and degree of distress associated with seven common heart failure symptoms: daytime dyspnea, orthopnea, fatigue, chest pain, edema, sleep problems, and dizziness or lightheadedness. Each symptom is rated using 4-point Likert-type response options. A response of "0" indicates absence of the symptom. When a symptom is present, patients rate symptom frequency (1 = less than once per week to 4 = nearly every day), severity (1 = mild to 4 = very severe), and symptom-related distress (1 = almost none to 4 = very much). Scores for each symptom are calculated by summing frequency, severity, and distress ratings. Total scores range from 0 to 84, with higher scores indicating greater symptom severity.
Mean Score on the Minnesota Living with Heart Failure Questionnaire (Quality of Life) | At baseline, 1 month, 3 months, and 6 months
  Quality of life will be assessed using the Minnesota Living with Heart Failure Questionnaire, developed by Rector et al. (1992). The questionnaire consists of 21 items evaluating the impact of heart failure on patients' physical, emotional, and social functioning, including symptoms such as dyspnea, peripheral edema, fatigue, anxiety, and depressive symptoms. Eight items assess the physical dimension (score range: 0-40), and five items assess the emotional dimension (score range: 0-25); the remaining items contribute to the total score only. Each item is scored on a 6-point Likert scale ranging from 0 ("no impact") to 5 ("very much"). Total scores range from 0 to 105, with lower scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in the primary and secondary outcome analyses, including outcome measure scores and relevant baseline characteristics.
Supporting Information: Study Protocol
Time Frame: Beginning after publication of the primary results and available upon reasonable request.
Access Criteria: Researchers who provide a methodologically sound proposal and agree to the terms of a data use agreement. Requests will be reviewed by the principal investigator. Access will be provided for academic, non-commercial research purposes only.

REFERENCES:
- [Background] Veroff DR, Sullivan LA, Shoptaw EJ, Venator B, Ochoa-Arvelo T, Baxter JR, Manocchia M, Wennberg D. Improving self-care for heart failure for seniors: the impact of video and written education and decision aids. Popul Health Manag. 2012 Feb;15(1):37-45. doi: 10.1089/pop.2011.0019. Epub 2011 Oct 17. PMID 22004181